CLINICAL TRIAL: NCT02676024
Title: Consolidating Tools for Outcomes in Resuscitation (CONTOUR)
Brief Title: Consolidating Tools for Outcomes in Resuscitation
Acronym: CONTOUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); University of Ottawa (Other); Children's Hospital of Eastern Ontario (Other); The Hospital for Sick Children (Other); Montreal Children's Hospital of the MUHC (Other); Alberta Children's Hospital (Other); Stollery Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20150075-01H
Record Dates: First submitted 2015-12-08; First posted 2016-02-05 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest; Cardiopulmonary Resuscitation; Simulation; Education
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Resuscitation teams will participate in a simulated pediatric cardiac arrest scenario, and provide standard CPR without being provided cognitive aids. Participants in this group will be allowed to use any cognitive aid that they happen to keep with them and would normally use in their practice, for example, flash cards or smart phone apps.
- Knowledge-based cognitive aid (Experimental): Resuscitation teams participate in a simulated pediatric cardiac arrest scenario, and provide standard CPR. However, they will be trained in using a knowledge-based cognitive aid, which will be used by a dedicated team member (the cognitive aid "reader").
  Interventions: Device: Knowledge-based cognitive aid
- Cognitive aids with roles defined (CARD) (Experimental): Resuscitation teams participate in a simulated pediatric cardiac arrest scenario, and provide standard CPR. Participants will be trained to use the cognitive aids with roles defined (CARD) system. However, they will not be given knowledge-based cognitive aids and there will be no dedicated cognitive aid reader in the team.
  Interventions: Device: Cognitive aids with roles defined (CARD)
- Integrated cognitive aids (Experimental): Participants will be trained to use the cognitive aids with roles defined (CARD) system and also in the use of a protocol-based cognitive aid, which will be used by a dedicated cognitive aid reader.
  Interventions: Device: Integrated cognitive aids

INTERVENTIONS:
Device: Knowledge-based cognitive aid — Trained on the use of a knowledge-based cognitive aid for pediatric cardiac arrests. Will be used by a dedicated team member (cognitive aid "reader").
  Arms: Knowledge-based cognitive aid
Device: Cognitive aids with roles defined (CARD) — Trained on the use of the cognitive aids with roles defined (CARD) system for pediatric cardiac arrests. Participants are given large identification cards to be worn, which enable the code leader to quickly recognize the individuals' purpose at the code. The card identifies specific tasks associated with the role, ensuring that the participant knows exactly what their task is. Will not have a dedicated team member during the scenario (cognitive aid "reader").
  Arms: Cognitive aids with roles defined (CARD)
Device: Integrated cognitive aids — Trained on the use of the cognitive aids with roles defined (CARD) system and also in the use of a protocol-based cognitive aid for pediatric cardiac arrests which will be used by a dedicated cognitive aid "reader".
  Arms: Integrated cognitive aids

SUMMARY:
In-hospital pediatric cardiac arrest is an important public health problem affecting almost 6000 children a year in the United States. As many as 3% of patients admitted to a children's hospital require cardiopulmonary resuscitation (CPR). Only a minority of children survive, of which around 35% go on to have a poor neurological outcome. International consensus guidelines on science and treatment recommendations for the management of pediatric resuscitation have existed for decades and are revised periodically by the International Liaison Committee on Resuscitation (ILCOR) based on available evidence. This consensus is then used by national councils such as the American Heart Association (AHA) and the Heart and Stroke Foundation of Canada (HSFC) to make guidelines for care. These guidelines focus on a structured approach to resuscitation, which emphasizes the rapid implementation of key interventions such as starting chest compressions, administering epinephrine and defibrillation. The goal of this study is to improve outcomes after cardiac arrest in children by improving adherence to consensus guidelines. The investigators aim to achieve this by conducting a multi-center, prospective, factorial randomized study with participating sites from the International Network for Simulation-based Pediatric Innovation, Research and Education (INSPIRE).

The specific aims of this study are to:

1. To evaluate the effectiveness of knowledge-based cognitive aids, namely the Pediatric Advanced Life Support (PALS) algorithm cards, in healthcare teams.
2. To evaluate the effectiveness of teamwork-based cognitive aids, namely the Cognitive Aids with Roles Defined (CARD) system, in healthcare teams.
3. To determine if there is a synergistic effect when adding the CARD system to the use of knowledge-based cognitive aids or indeed whether using both these tools together has unintended consequences and reduces the added value of each technique.
4. To identify whether additional simulation-based team training in the use of cognitive aids results in a significant improvement in performance over an e-learning module.

The investigators hypothesize that (i) knowledge-based cognitive aids will significantly improve the performance of healthcare teams in providing PALS in a simulated setting, (ii) that teamwork-based cognitive aids (CARD) will significantly improve the performance of healthcare teams in providing PALS in a simulated setting, and that (iii) adding the CARD system to knowledge-based aids will have an added and synergistic effect, (iv) that the team performance in all study arms will improve after simulation based training, but that the groups with cognitive aids will continue to out-perform the groups without cognitive aids.

DETAILED DESCRIPTION:
This study utilizes a prospective, randomized controlled, factorial study design, which examines the effect of integrating different elements of cognitive aids for training pediatric resuscitation team members. Recruited participants will be asked to perform as members of a multi-professional pediatric resuscitation team. The study uses simulation-based training as the primary method to evaluate the effect of both knowledge- and team-based cognitive aids on team performance, as measured by adherence to PALS guidelines. Participants will be teams of multi-professional pediatric resuscitation healthcare providers (physician, registered nurse, registered respiratory therapist). All participants will undertake a pre-test scenario, without access to either cognitive aid, regardless of group allocation. Participants will then be randomized to one of the four study arms using a list generated by an independent statistician. Randomization will be stratified by institution so that there are equal numbers of teams in each study arm in each participating institution of the multi-center study.

In study arm 1 (control), resuscitation teams will participate in a simulated pediatric cardiac arrest scenario, and provide standard CPR without being provided cognitive aids. Participants in this group will be allowed to use any cognitive aid that they happen to keep with them and would normally use in their practice, for example, flash cards or smart phone apps. In study arm 2 (knowledge-aid), resuscitation teams will participate in the same scenario without using the CARD system but will be trained in the use of a knowledge-based cognitive aid, which will be used by a dedicated team member (the cognitive aid "reader"). In study arm 3 (CARD), participants will be trained to use the cognitive aids with roles defined (CARD) system but will not be given knowledge-based cognitive aids and there will be no dedicated cognitive aid reader in the team. In study arm 4 (integrated cognitive aid), participants will be trained to use the CARD system and also in the use of a protocol-based cognitive aid, which will be used by a dedicated cognitive aid reader.

All groups will then undertake a 20-minute e-learning module. E-learning modules will be developed to illustrate the principles of crisis resource management using text, images and short videos (of simulated scenarios) illustrating high- and low- performance in leadership, teamwork and task management. For the control group, the content will focus on team training principles and the PALS algorithm. For the knowledge-aid group, the content will also focus on team training principles and the PALS algorithm adding an introduction of the principle of using the knowledge-based cognitive aids provided with a cognitive aid "reader" designated by the team leader who will use a "do-verify" approach to the cognitive aid. For the CARD group, the content will also focus on team training principles and the PALS algorithm adding an introduction of the principles of the CARD system. For the integrated cognitive aid group, the content will focus on team training principles and the PALS algorithm adding an introduction of the principles of the CARD system and the principle of using the knowledge-based cognitive aids provided with a cognitive aid "reader" designated by the team leader who will use a "do-verify" approach to the cognitive aid.

All participants will then undergo a post-test scenario, with cognitive aids provided as per group allocation. A debriefing will follow in order to delineate the additional effect of simulation-based learning on the e-module. All study arms will then undertake a second-post-test scenario, with cognitive aids related to their group allocation followed by a second debriefing. Participants will be asked to complete a demographic questionnaire and a questionnaire on the use of cognitive aids.

In order to standardize scenarios between sites, the investigators will script the content of each scenario, including set transitions from one clinical state to another, programmed responses to expected interventions, and a pre-set duration. The scenarios will be piloted at the main study site and videos circulated to all other sites before piloting at those locations.

Scenario for assessment (pre-test, post-test 1 and post-test 2)

One 12-minute pediatric cardiac arrest resuscitation scenario will be developed to address PALS-based cognitive and clinical performance, as well as compliance with American Heart Association guidelines. This scenario has two phases: the first being a non-shockable rhythm arrest (six minutes) and the second being a shockable rhythm arrest (six minutes). The case history before the arrest and the exact rhythms will be different in each phase to prevent over familiarity with the scenarios but the expected management of the arrest is the same in each to minimize variations in difficulty of scenario from pre-test to post-test:

1. Pre-test: bronchiolitis; pulseless electrical activity/ventricular fibrillation
2. Post-test 1: sepsis, pulseless electrical activity/ventricular tachycardia
3. Post-test 2: myocarditis; pulseless activity/ventricular tachycardia

The scenario is designed to test clinical performance during both cardiac arrest algorithms. To ensure consistency in delivery of the scenario between recruitment sites, each site will be provided with a pre-programmed scenario and a script for the simulation facilitator, outlining specifically how to run the scenario, how to introduce the patient, and how/when to provide verbal cues to the resuscitation team. During a pre-study run-in phase, each recruitment center will have to conduct and transmit 2 successful case scenarios using this format to the research coordinating center. This will allow the investigators to confirm adequate quality of audiovisual content and sound before the site is allowed to conduct and submit data from their site. Videos and data collected during the run-in phase will not be analyzed for inclusion in the main study. Participants recruited during this phase will not be eligible for inclusion in the study.

All recruitment sites will utilize the same make/brand of pediatric simulator for this study. The Laerdal SimBaby is widely used across Canada and the Unites States and is capable of reproducing physiological responses to medical interventions. This simulator is connected to a monitor where vital signs (heart rhythm, respiratory rate, oxygen saturation, blood pressure, temperature) are displayed. Through a computer interface, an operator can run pre-programmed scenarios where vital signs on the monitor and physical findings on the simulator change in real time. The mannequin is capable of producing heart sounds, breath sounds and palpable pulses. The simulator can be bag-mask ventilated, the trachea intubated and the heart defibrillated. Our cardiac arrest scenario will be pre-programmed into the simulator to ensure consistency between recruitment sites and study groups. The investigators will ensure as much standardization as possible between centers in the physical environment for the scenario, including the same availability and location of equipment, including a similar sized room.

Video rating will be by multiple independent raters with expertise in both simulation and pediatric resuscitation, who will be blinded to the research question. Raters will be trained in the use of the assessment tools by the primary investigator and co-investigators using video conferencing technology. The rater training process will consist of (i) a short tutorial on how to use the rating tools, (ii) each rater independently rating similar scenarios to those used in the study (which will not be used in the analysis), (iii) a group discussion of the ratings led by the principle investigator in order to resolve differences and obtain consensus. Approximately 10% of the videos will be rated in duplicate in order to establish inter-rater reliability.

ELIGIBILITY:
Inclusion Criteria:

Team Leader: Resident in Pediatrics, Anesthesia, or Emergency Medicine training programs and College of Family Physicians of Canada resident. Fellows in Pediatric Emergency Medicine, Pediatric Critical Care or Pediatric Anesthesia sub-specialty training programs. Staff general Pediatricians.

Team members: Registered Nurses, Respiratory Therapists, Pediatric Residents.

Exclusion Criteria:

Decline to consent to participation. Those that would not attend a code outside of the operating room.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Estimated)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to PALS guidelines as measured by the clinical performance tool (CPT) | At baseline (pre-test)
  Simulated scenarios will be videotaped. These will be scored according to the CPT which is a task-specific checklist that is reliable and validated in assessing performance in a multi-professional team
Adherence to PALS guidelines as measured by the clinical performance tool (CPT) | At post-test 1 (same day as pre-test)
  Simulated scenarios will be videotaped. These will be scored according to the CPT which is a task-specific checklist that is reliable and validated in assessing performance in a multi-professional team
Adherence to PALS guidelines as measured by the clinical performance tool (CPT) | At post-test 2 (same day as pre-test)
  Simulated scenarios will be videotaped. These will be scored according to the CPT which is a task-specific checklist that is reliable and validated in assessing performance in a multi-professional team

SECONDARY OUTCOMES:
Time to initiation of cardiopulmonary resuscitation | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped and timing will be measured by the video raters.
Time to administration of epinephrine | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped and timing will be measured by the video raters.
Time to defibrillation after the start of phase 2 of the scenario (VF) | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped and timing will be measured by the trained video raters.
Percentage of "no-flow" time without chest compressions | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped and timing will be measured by the video raters.
Team Emergency Assessment Measure (TEAM) scale | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped. Videos will be scored by trained raters according to the validated TEAM scale.
Frequency of use of the knowledge-based cognitive aid | This outcome measure will be assessed during the pre-test, post-test 1 and post-test 2. All the scenarios take place on the same day.
  Simulated scenarios will be videotaped. Frequency of use of the knowledge-based cognitive aid will be measured by trained raters using an anchored 7-point Likert scale

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario